CLINICAL TRIAL: NCT07103720
Title: The Nonirritating Concentrations of Midazolam, Ketamine, and Ondansetron
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Arizona Biomedical Research Commission (ABRC) (Other)
Responsible Party: Principal Investigator, Alexei Gonzalez-Estrada, MD, Alexei Gonzalez-Estrada, M.D., Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 25-001858
Record Dates: First submitted 2025-07-27; First posted 2025-08-05 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity | interventions — Skin Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Group (Experimental): Study team is developing a new diagnostic skin testing procedure to determine non-irritant concentrations of midazolam, ketamine and ondansetron administered to patients before, during or after surgery.
  Interventions: Diagnostic Test: Skin Testing

INTERVENTIONS:
Diagnostic Test: Skin Testing — Participants will undergo skin prick testing and intradermal test injections at 5 increasing concentrations of midazolam, ketamine and/or ondansetron during one single study visit.

SUMMARY:
Perioperative anaphylaxis is a potentially life-threatening drug allergic reaction that can occur during anesthetic procedures. The purpose of this research is to determine the maximal nonirritating skin testing concentrations of midazolam, ketamine and ondansetron. These drugs are FDA approved and commonly used before, during and after surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Not have a history of an adverse reactions to midazolam, ketamine or ondansetron
* Ability to understand study procedures and to comply with them for the entire length of the study.
* Contraception is not necessary, and we will include women of reproductive capability.

Exclusion Criteria:

* Unstable patients.
* History of any adverse reaction (allergy or sensitivity) to midazolam, ketamine or ondansetron.
* Pregnant and Pediatric patients
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Nonirritating Concentrations of Midazolam, Ketamine, and Ondansetron. | 1 Day
  Determine the maximal nonirritating concentrations of midazolam, ketamine and ondansetron

SECONDARY OUTCOMES:
Skin Testing Results | 1 Day
  Determine the frequency of false positive test results in patients who have received Midazolam, Ketamine or Ondansetron in the past.

CONTACTS AND LOCATIONS:
Overall Officials: Alexei Gonzalez Estrada, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials